CLINICAL TRIAL: NCT00941369
Title: Health Assessment, Patient Treatment Satisfaction and Quality-of-Life in Insulin-naive Type 2 Diabetes Patients Uncontrolled on Oral Hypoglycemic Agent Treatment Initiating Basal Insulin Therapy With Either Insulin Glargine or NPH Insulin
Brief Title: Health Assessment, Patient Treatment Satisfaction and Quality-of-Life in Insulin-Naive Type 2 Diabetes Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_04079; 2009-019013-59(EudraCT)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (2):
- 1 (Experimental): Insulin glargine: Lantus® (100 U/ml) in TactiPen® re-usable pen
  Interventions: Drug: Insulin Glargine (HOE901)/NPH Insulin
- 2 (Active Comparator): Neutral Protamine Hagedorn basal insulin: Insuman® Basal (100 I.U./ml) in TactiPen® re-usable pen
  Interventions: Drug: Insulin Glargine (HOE901)/NPH Insulin

INTERVENTIONS:
Drug: Insulin Glargine (HOE901)/NPH Insulin — Arm 1: Subcutaneous injection of Insulin Glargine with the TactiPen® injector pen once daily at any time, but each day at the same time
  Arm 2: Subcutaneous injection of Protamine Hagedorn basal insulin with the TactiPen® injector pen once or twice daily at the discretion of the treating physician
  The starting dose is 10 I.U. (NPH basal insulin) resp. 10 U (insulin glargine) per day.
  The dose adjustments will be based on the results of self-monitoring.

SUMMARY:
Primary Objective:

To investigate the impact of insulin glargine versus Neutral Protamine Hagedorn basal insulin on a composite diabetes related quality of life score (DRQoL).

Secondary Objective:

A comparison of combination therapy with insulin glargine versus Neutral Protamine Hagedorn basal insulin from baseline to endpoint in terms of:

* Glycaemic parameters: 7 blood glucose profiles
* Incidence of confirmed symptomatic hypoglycemia as well as confirmed severe hypoglycemia
* Change in lipid status

ELIGIBILITY:
Inclusion criteria:

* Patients with type 2 diabetes mellitus (no history of ketoacidosis) according to ADA criteria.
* Treatment with a combination of maximum 2 substance classes on a stable dosage during the last 3 months: metformin and/or sulfonylurea.
* No pre-treatment with any insulin in the last 3 months before the study.
* Glycated Haemoglobin A1c (HbA1c) value between > or = 7.0 and > or = 9.5%
* Fasting Blood Glucose (FBG) > or = 120 mg/dl (6.7 mmol/l).
* Body mass index < 40 kg/m.
* Ability to read and understand German language.
* Ability and willingness to follow a tight antidiabetic therapy and to perform blood glucose self monitoring on a regular basis.
* Women of childbearing potential who will take adequate contraceptive protection.

Exclusion criteria:

* Patients with type 1 diabetes mellitus.
* Any history of ketoacidosis.
* Pregnancy.
* Prior treatment with insulin.
* Treatment with more than two oral agents within the last 3 months or continuous treatment with thiazolidinediones, GLP-1 receptor agonists or with Dipeptidyl-Peptidase IV (DPP-IV) inhibitors.
* History of drug or alcohol abuse.
* Diabetic retinopathy with surgical treatment (laser photocoagulation or vitrectomy) in the last 3 months prior to study entry or which may require surgical treatment within 3 months of study entry.
* Following pancreatectomy.
* Impaired hepatic function.
* Impaired renal function.
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
* Evidence of an uncooperative attitude, including poor compliance to any (antidiabetic) treatment.
* Inability to attend follow-up visits.
* Current treatment because of a mental disorder according to ICD 10(F 5 Diagnoses).
* Patients that are in a relationship of dependance with the investigator(s) and/or the sponsor.
* Systemic corticoids > 7,5 mg prednisolon equivalent or <or=7,5 mg prednisolon equivalent for less than 2 months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Health Assessment, Patient treatment satisfaction and Quality-of-Life | At baseline (visit 2: randomization), at 24 weeks after the randomization (visit 7: cross over visit) and 48 weeks after the randomization (visit 12: endpoint)

SECONDARY OUTCOMES:
Glycaemic parameters assessment | At baseline (visit 2: randomization), 24 weeks after the randomization (visit 7) and 48 weeks after the randomization (visit 12: endpoint)
Anteropometric data (Weight, waist circumference) assessment | At baseline (visit 2: randomization), 24 weeks after the randomization (visit 7) and 48 weeks after the randomization (visit 12: endpoint)
Lipid assessment | At 24 weeks after the randomization (visit 7) and 48 weeks after the randomization (visit 12: endpoint)
Hypoglycemia assessment | Throughout the study from starting until the week 48

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Riederer, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Berlin, Germany

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- [Derived] Hermanns N, Kulzer B, Kohlmann T, Jacob S, Landgraf W, Theobald K, Haak T. Treatment satisfaction and quality-of-life between type 2 diabetes patients initiating long- vs. intermediate-acting basal insulin therapy in combination with oral hypoglycemic agents--a randomized, prospective, crossover, open clinical trial. Health Qual Life Outcomes. 2015 Jun 9;13:77. doi: 10.1186/s12955-015-0279-4. PMID 26055391